CLINICAL TRIAL: NCT01429285
Title: Safety and Efficacy of Intravenous Hydromorphone Using Incremental Doses of 0.5 mg in Elderly ED Patients With Acute Severe Pain
Brief Title: Safety and Efficacy of Intravenous Hydromorphone in Elderly Emergency Department Patients With Acute Severe Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, Prinicipal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMC 08-11-387
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: Pain; Hydromorphone; Acute; Emergency Department
MeSH Terms: conditions — Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydromorphone (Experimental): Hydromorphone protocol
  Interventions: Drug: Hydromorphone
- Usual care (Active Comparator): Usual care
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: Hydromorphone — 0.5 mg IV hydromorphone followed by an optional 0.5 mg IV dose
  Other Names: Dilaudid
  Arms: Hydromorphone
Drug: Usual care — Attending administers any IV opioid in any dose he chooses
  Arms: Usual care

SUMMARY:
The hydromorphone protocol is more effective than usual care in Emergency Department (ED) patients age 65 years and older in terms of proportion who choose to forgo additional pain medication within 60 minutes post-baseline in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 65 years: This is a study of elderly patients.
2. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in Emergency Department (ED) literature.
3. ED attending physician's judgment that patient's pain may warrant intravenous (IV) opioids: The factors that influence the decision to use parenteral opioids are complex and extensive. An approach that is commonly taken to address the issue of patient selection in drug trials is to use a specific condition (e.g., renal colic) or treatment (e.g., post-hysterectomy) that would generally be thought to be appropriately treated with an opioid analgesic, thereby eliminating individual judgment about eligibility for the study. However in order to assess the role of opioids with the widest generalizability in the ED setting, the investigators decided to enroll patients with a variety of diagnoses, all with a complaint of acute pain. Opioids are not an appropriate treatment for all patients who present with a complaint of pain (e.g., gastroenteritis, migraine). Therefore, unless there is a restriction to patients with a specific diagnosis, either a comprehensive list of diagnoses and situations in which opioids are indicated must be specified, or clinical judgment needs to be used. The investigators have opted for the latter alternative.
4. Normal mental status: In order to provide measures of pain experienced the patient needs to have a normal mental status. The investigators will use a 6-item screener (Wilber 2008) as an indicator of sufficiently normal mental status to participate in the study.

Exclusion Criteria:

1. Prior use of methadone: the effect of methadone use on the perception of acute pain is unknown and suspected to be altered. The investigators feel that the needs of patients on methadone may exceed the dosage ceiling of 1 mg that will be used for this study. Similar to sickle cell patients and chronic cancer patients, patients on methadone usually require significantly higher doses of opioids to control their pain. Thus, the investigators feel that it would be unethical to restrict the dose that this subset of patients can receive.
2. Use of other opioids or tramadol within past seven days: to avoid introducing bias related to opioid tolerance that may alter the response to the study medication thereby masking the medication's effect.
3. Prior adverse reaction to opioids.
4. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in alteration in pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, migraine, and peripheral neuropathies.
5. Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter perception, report, and treatment of pain.
6. Systolic blood pressure <90 mm Hg: Opioids can produce peripheral vasodilation that may result in orthostatic hypotension.
7. Oxygen saturation <95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
8. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
9. C02 measurement greater than 46: In accordance with a similar study (04-12-360), three subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46, then the patient will be excluded from the study. The 3 subsets are as follows:

   * All patients who have a history of chronic obstructive pulmonary disease (COPD)
   * All patients who report a history of asthma together with greater than a 20 pack-year smoking history
   * All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Emergency Department, The Bronx, New York, United States

REFERENCES:
- [Derived] Chang AK, Bijur PE, Davitt M, Gallagher EJ. Randomized clinical trial of an intravenous hydromorphone titration protocol versus usual care for management of acute pain in older emergency department patients. Drugs Aging. 2013 Sep;30(9):747-54. doi: 10.1007/s40266-013-0103-y. PMID 23846749

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydromorphone | Usual Care
Started | 175 | 175
Given IV Opioids | 166 (9 patients never given IV opioids) | 171 (4 patients never given IV opioids)
Completed Primary Outcome Data | 161 (5 patients had missing data) | 168 (3 patients had missing data)
Confirmation of no Duplicate Enrollment | 153 (8 patients were enrolled twice at two separate ED visits, which was only noted at study conclusion.) | 166 (2 patients were enrolled twice, at two separate ED visits, which was only noted at study conclusion)
Completed | 153 | 166
Not Completed | 22 | 9
Not completed — Protocol Violation | 9 | 4
Not completed — Missing Data | 5 | 3
Not completed — Erroneously Enrolled Twice | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone | Usual Care | Total
Number analyzed (Participants) | 153 | 166 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (7) | 74 (6) | 74 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 108 | 213
  Male | 48 | 58 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 97 | 103 | 200
  African American | 35 | 44 | 79
  White | 15 | 16 | 31
  Other | 6 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 153 | 166 | 319
Weight [Mean (Standard Deviation); unit: lbs] | 162 (33) | 165 (38) | 164 (36)
Diagnosis [Count of Participants; unit: Participants]
  Non-specific abdominal pain | 50 | 57 | 107
  Musculoskeletal pain | 24 | 24 | 48
  Back pain | 14 | 13 | 27
  Colitis/diverticulitis | 14 | 10 | 24
  Small Bowel Obstruction | 12 | 13 | 25
  Extremity fracture | 11 | 7 | 18
  biliary colic/cholecystitis | 6 | 11 | 17
  Kidney stone/pyelonephritis | 7 | 11 | 18
  Appendicitis | 0 | 6 | 6
  Other (pancreatitis, perforated viscus, etc) | 15 | 14 | 29
Pain Intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS), with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable").
  Participants
    NRS = 3-6 | 12 | 13 | 25
    NRS = 7 | 14 | 20 | 34
    NRS = 8 | 31 | 28 | 59
    NRS = 9 | 20 | 24 | 44
    NRS = 10 | 76 | 81 | 157
Nauseated or vomited before receiving opioids in the ED [Count of Participants; unit: Participants]
  Yes | 65 | 77 | 142
  No | 87 | 89 | 176
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Treatment
Description: Number of patients with "successful treatment" is defined as the number of patients who declined additional pain medication within 1 hour of study entry when asked the question, "Do you want more pain medication?". This measure looks at declining pain medication at either 15 minutes or 60 minutes, whereas 4. Post-Hoc refers only to the answer to the question at the 60 minute mark post-baseline.
Time Frame: 1 hour
Population: The discrepancy between the number of patients enrolled and randomized and the number analyzed is due to patient never being given IV opioids (13), enrolled twice (10), and missing primary outcome data (8)
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
Participants
  Achieved satisfactory analgesia within 60 min | 127 | 137
  No satisfactory analgesia within 60 min | 26 | 29

2. Secondary Outcome: Mean Change in Pain Intensity From Baseline to 60 Minutes
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable"). The change in scores over time is calculated by subtracting the score at 60 minutes from the score at baseline (before treatment). These change values were then averaged.
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
units on a scale | 5.4 (2.9) | 5.2 (3.1)

3. Post Hoc Outcome: Number of Patients Who Achieved Satisfactory Analgesia at 15 Minutes Post-baseline
Description: Satisfactory Analgesia is defined as declining additional pain medication when asked the question, "Do you want more pain medication?"
Time Frame: 15 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
Participants | 89 | 111

4. Post Hoc Outcome: Number of Patients Who Achieved Satisfactory Analgesia at 60 Minutes Post-baseline
Description: "Satisfactory analgesia" is defined as the patient declining additional pain medication when asked the question, "Do you want more pain medication?". This measure refers only to the answer to this question asked at the 60 minute mark. The Primary Outcome (1. Primary Outcome - Number of Patients with successful treatment) refers to the answering "no" to this question at 15 minutes or 60 minutes post-baseline.
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
Participants | 111 | 119

5. Post Hoc Outcome: Number of Patients With 50% or Greater Decline in Pain Intensity Score From Baseline to 60 Minutes
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable"). The 50% or greater change in pain score is measured by subtracting the pain score at 60 minutes from the pain score at baseline, then dividing that value by the original baseline value and multiplying by 100% to get a percent change value.
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
Participants | 106 | 107

6. Post Hoc Outcome: Number of Patients With a Pain Intensity Score of 3 or Less at 60 Minutes
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable").
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
Participants | 83 | 87

7. Post Hoc Outcome: Pain Intensity Score at 60 Minutes
Description: as for outcome 6
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 153 | 166
units on a scale | 3 [0 to 5] | 3 [0 to 6]

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: The discrepancy between the number of patients enrolled and randomized and the number analyzed is due to patient never being given IV opioids (13), enrolled twice (10), and missing primary outcome data (8)
Arm/Group | Hydromorphone | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/166
Other Adverse Events (participants affected / at risk) | 27/153 | 32/166
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Hydromorphone (N=153) | Usual Care (N=166)
Oxygen saturation <95% (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Systolic blood pressure <90 mmHg (Vascular disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 8
Nausea (Gastrointestinal disorders) | 10/87 | 6/89 — excluding patients who were nauseated or vomiting before receiving initial IV opioids
Vomiting (Gastrointestinal disorders) | 4/87 | 3/89 — excluding patients who were nauseated or vomiting before receiving initial intravenous opioid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes